CLINICAL TRIAL: NCT06879821
Title: Effectiveness of a High-intensity Functional Training (HIFT) Program on Functional and Cognitive Performance in People with Parkinson's Disease.
Brief Title: High-intensity Functional Training on Functional and Cognitive Performance in People with Parkinson's Disease.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Para La Investigacion Hospital La Fe (Other)
Responsible Party: Principal Investigator, Marta Aguilar-Rodriguez, Assistant Professor, University of Valencia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2022_TesisIVargas_UV
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups: experimental group (EG) and control group (CG). The experimental group will perform a HIFT training program and the control group will follow their routine of physical and cognitive exercises, which will be recorded for control purposes.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The experimental group will perform a high-intensity functional training program twice a week for 10 weeks.
  Interventions: Other: high intensity functional training
- Control Group (No Intervention): The control group will continue to carry out their physical and cognitive exercise routine during the week, recording their activity in days and sessions.

INTERVENTIONS:
Other: high intensity functional training — The pillar of rehabilitation will be based on high intensity functional training. 45-minute sessions divided into 5 minutes of warm-up, 35 minutes of functional exercises, and 5 minutes of going back to bed and cooling down. The 35 minutes of exercises were divided into 3 categories: lower extremity exercises, upper extremity exercises, and static and dynamic coordination and balance exercises. Each category will consist of 3 exercises per session, performing 2-3 series with a maximum of repetitions of 10-RM. The progression of the load will be progressively increased in weeks 3, 5 and 8 between 40-60% of the 1-RM.
  Other Names: HIFT
  Arms: Experimental group

SUMMARY:
Parkinson's disease (PD) is a progressive and chronic neurodegenerative disease, which presents signs and symptoms both motor (impaired gait, posture, balance, etc.) and cognitive (memory loss, dementia, etc.), all of which are causing disability and assuming a high economic cost. Currently, there are already certain authors who have shown how a high-intensity interval training (HIIT) protocol produces improvements in cognitive and physical performance in healthy adults6 and in people with multiple sclerosis. However, another modality has been created, such as high-intensity functional training (HIFT), which can benefit different populations, both healthy and pathological, due to the multimodal nature of the exercises. Thanks to multimodality, more aspects such as agility, coordination and precision of movements are worked on compared to unimodal HIIT programs that make this relevant work difficult in a person's daily life. The current study aims to demonstrate the effectiveness of a HIFT training protocol in a specific population, such as people with Parkinson's disease.

DETAILED DESCRIPTION:
The hypothesis is that high-intensity functional training (HIFT), at a motor and cognitive level, provides a greater benefit than conventional programs of strength, balance and cognition, on the functionality and cognitive capacity of people with Parkinson's disease.

Overall objective:

- To assess whether the HIFT training program is associated with significant improvements in functional and cognitive capacity compared to conventional strength, balance and cognition programs in Parkinson's patients.

Secondary objectives:

1. To assess whether the HIFT program improves the quality of life in patients with PD.
2. To study whether the HIFT program reduces the degree of dependency of patients with PD.
3. To determine if the HIFT program improves physical performance in patients with PD
4. To assess whether the HIFT program reduces the risk of falls in patients with PD.
5. To investigate whether the HIFT program improves balance in patients with PD.
6. To determine if the HIFT program improves functional capacity in patients with PD.
7. To study whether the HIFT program improves cognitive function in patients with PD

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease.
* Stage I or II (Hoehn - Yahr Scale).
* Age between 45 and 80 years.
* Independent ambulation for 10 consecutive minutes.
* Regular physical exercise.

Exclusion Criteria:

* Medical contraindication for physical activity, deafness or limited hearing and very low vision or blind.
* Vestibular disorders that compromise balance.
* Psychotic or severe cognitive disorder.
* Decompensation or changes in medication.
* Surgical intervention in the last 6 months.
* Sedentary persons

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Short physical performance battery (SSPB) | 10 minutes
  Functional performance evaluation.
Trail Making Test A y B | 15 minutes
  Evaluation of visual search, scanning, processing speed, mental flexibility and executive functions.

SECONDARY OUTCOMES:
SF-12 Health Questionnaire | 10 minutes
  Assessing Perceived Quality of Life
Barthel index | 10 minutes
  Evaluation of the degree of dependence in activities of daily living.
fall risk assessment scale | 5 minutes
  Fall Risk Assessment
2-minute walk test (2-MWT) | 5 minutes
  Evaluation of functional capacity
Mini Mental State Examination | 20 minutes
  Assessment of cognitive function

OTHER OUTCOMES:
The Borg Scale | 2 minutes
  Rating of perceived exertion

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No